CLINICAL TRIAL: NCT02968420
Title: Long Term Immune Memory Responses to Human Papillomavirus (HPV) Vaccination Following 2 Verses 3 Doses of Quadrivalent HPV Vaccine
Brief Title: Long Term Immune Memory Responses to HPV Vaccination Following 2 vs 3 Doses of Quad-HPV Vaccine
Acronym: Merck08
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Principal Investigator, Manish Sadarangani, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-00700
Record Dates: First submitted 2016-08-19; First posted 2016-11-18 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Human Papillomavirus
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Group 1: girls who received 2 doses of Q-HPV vaccine at 0, 6 month schedule 8-10 years ago when they were between 9-13 years of age at the time of the first dose. The intervention of a single dose of licensed Gardasil 9 vaccine (Human Papillomavirus 9-valent Vaccine, Recombinant) will be administered at Day 0 of the study.
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant
- Group 2 (Active Comparator): Group 2: girls who received 3 doses of Q-HPV vaccine at 0, 2, 6 month schedule 8-10 years ago when they were between 9-13 years of age at the time of the first dose. The intervention of a single dose of licensed Gardasil 9 vaccine (Human Papillomavirus 9-valent Vaccine, Recombinant) will be administered at Day 0 of the study.
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant
- Group 3 (Active Comparator): Group 3: young women who received 3 doses of Q-HPV vaccine at 0, 2, 6 month schedule 8-10 years ago when they were between 16-26 years of age at the time of the first dose. The intervention of a single dose of licensed Gardasil 9 vaccine (Human Papillomavirus 9-valent Vaccine, Recombinant) will be administered at Day 0 of the study.
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant

INTERVENTIONS:
Biological: Human Papillomavirus 9-valent Vaccine, Recombinant — All groups will receive a single dose of the Gardasil9 vaccine at Visit 1/Day 0 of the study.
  Other Names: Gardasil9

SUMMARY:
The overall aim of this study is to further understand the memory response to HPV vaccination in subjects who have received 2 versus 3 doses of quadrivalent HPV vaccine. Although memory responses can be detected shortly after immunization, the best approach to measure the long-lasting anamnestic response is to challenge with a booster dose years (> 5) after the original exposure.

DETAILED DESCRIPTION:
This is a single center, interventional study to evaluate long term memory response to Q-HPV vaccination and to natural infection. Memory response will be assessed by measuring seroprotection 8-10 years post Q-HPV vaccination and to challenge with a booster dose years after the original exposure to measure the long-lasting anamnestic response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the participant.
* Participant whom the investigator believes can and will comply with the requirements of the protocol.
* General good health.
* Immunized with Q-HPV vaccine between the ages of 9-13 or 16 to 26 years on the BCGov01 study or the BC provincial program.
* Participant who is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study. Examples of effective methods of birth control include:

  * Abstinence (no sexual activity)
  * Hormonal contraceptives including oral, injectable, implants & skin patches
  * Intrauterine device (IUD)
  * Male partner sterilization
  * Male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository)
  * Male condom combined with a female diaphragm, whether with or without a vaginal spermicide (foam, gel, cream, or suppository)
  * Adequate contraception does not apply to participants with same sex partners, when this is their preferred and usual lifestyle

Exclusion Criteria:

* Received more than 3 doses of Q-HPV vaccine
* Received any doses of HPV9 vaccine
* Systemic hypersensitivity to Q-HPV vaccine or HPV9 vaccine or severe reaction to any previous dose of Q-HPV vaccine.
* Receipt of blood or blood product within 3 months prior to Visit 1.
* Receipt of a live vaccine within 28 days or an inactive vaccine within 14 days of Visit 1
* Immune compromise resulting from disease or immunosuppressive systemic medication use within 3 months prior to Visit 1.
* Inadequate participant fluency in English to provide fully informed consent.
* Participant who is currently pregnant or planning a pregnancy during the course of the trial

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobi Kollmann, MD PhD, Principal Investigator — Vaccine Evaluation Center, University of British Columbia; Manish Sadarangani, BM BCh DPhil, Principal Investigator — Vaccine Evaluation Center, University of British Columbia
Locations (1):
- Vaccine Evaluation Center, BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
If IPD is required, please contact the study team for further discussions- any sharing will be dependent on alignment with original informed consent obtained from study participants and in agreement with the study team.

REFERENCES:
- [Background] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Derived] Carter JJ, Smith RA, Scherer EM, Skibinski DAG, Sankaranarayanan S, Luxembourg A, Kollmann T, Marty KD, Sadarangani M, Dobson S, Galloway DA. Term immune memory responses to human papillomavirus (HPV) vaccination following 2 versus 3 doses of HPV vaccine. Vaccine. 2025 Mar 19;50:126817. doi: 10.1016/j.vaccine.2025.126817. Epub 2025 Feb 5. PMID 39914257

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.05 (.89) | 21.95 (1.66) | 30.02 (3.34) | 24.67 (4.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 4 | 13
  Chinese | 0 | 0 | 1 | 1
  Other/mixed | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 6 | 18
Weight [Mean (Standard Deviation); unit: kg] | 74.60 (18.03) | 72.25 (26.51) | 73.75 (15.40) | 73.53 (19.31)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 27.37 (6.69) | 24.23 (6.15) | 25.63 (3.42) | 25.74 (5.42)

OUTCOME MEASURES:

1. Primary Outcome: B Memory Cell Response (% of Memory B Cells That Are Antigen-specific)
Description: To compare the B memory cell populations between girls that received either a primary 2 or 3 dose series, who are then challenged with a subsequent dose after 120 months
Time Frame: At Day 30 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Mean (Standard Deviation); unit: % of memory B cells that are Ag-specific
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
% of memory B cells that are Ag-specific
  HPV16 | 0.61 (0.49) | 0.94 (0.94) | 0.36 (0.23)
  HPV18 | 0.08 (0.18) | 0.11 (0.13) | 0.03 (0.05)

2. Primary Outcome: Plasmablast Response (% of All B Cells That Are Plasmablasts)
Description: To compare the plasmablast populations between girls that received either a primary 2 or 3 dose series, who are then challenged with a subsequent dose after 120 months
Time Frame: At Day 7 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Mean (Standard Deviation); unit: % of all B cells that are plasmablasts
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
% of all B cells that are plasmablasts | 2.37 (2.51) | 3.14 (3.53) | 5.37 (6.46)

3. Secondary Outcome: Variable Gene Usage (Comparison of the Nucleotide Sequences of Antigen-specific Antibody Heavy and Light Chain Variable Region Sequences)
Description: To compare the extent of somatic hypermutation and the variable gene usage between girls that received either a primary 2 or 3 dose series
Time Frame: At Day 7 and Day 30 post challenge dose of Human Papillomavirus 9-Valent vaccine
Population: The extent of somatic hypermutation was planned by comparing the nucleotide sequences of the heavy and light chain variable region sequences of each antibody cloned in this study to germ line sequences of these genes in public databases. This was not possible due to insufficient quality of DNA for sequencing.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Serum Antibody Response (cLIA) - Geometric Mean Titer
Description: To compare the serum antibody responses (cLIA) to HPV 6, 11, 16 & 18 at month 120 in females that received either a primary 2 or 3 dose series, who are then challenged with a subsequent dose
Time Frame: At Day 7 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
antibody titer
  HPV6 | 338 [111 to 1027] | 1864 [1411 to 2461] | 699 [129 to 3780]
  HPV11 | 1277 [592 to 2753] | 5071 [2361 to 10892] | 3807 [1096 to 13224]
  HPV16 | 4922 [1765 to 13731] | 15237 [6966 to 33328] | 10122 [3475 to 29481]
  HPV18 | 855 [461 to 1585] | 2140 [897 to 5105] | 807 [305 to 2134]

5. Secondary Outcome: Serum Antibody Response (cLIA) - Geometric Mean Titer
Description: as for outcome 4
Time Frame: At Day 30 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
antibody titer
  HPV6 | 1313 [376 to 4586] | 2722 [1472 to 5033] | 815 [135 to 4924]
  HPV11 | 3430 [1418 to 8299] | 6042 [3255 to 11214] | 5778 [2919 to 11439]
  HPV16 | 21135 [11337 to 39399] | 21768 [11797 to 40170] | 18930 [11126 to 32208]
  HPV18 | 3326 [1197 to 9245] | 2615 [1033 to 6620] | 1312 [676 to 2548]

6. Secondary Outcome: Serum Antibody Response (Total IgG) - Geometric Mean Titer
Description: To compare the serum antibody responses (total IgG) to HPV 6, 11, 16 & 18 at month 120 in females that received either a primary 2 or 3 dose series, who are then challenged with a subsequent dose
Time Frame: At Day 7 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
antibody titer
  HPV6 | 1263 [437 to 3650] | 6079 [3682 to 10036] | 3712 [1036 to 13302]
  HPV11 | 1009 [308 to 3306] | 5184 [2644 to 10164] | 3371 [947 to 11997]
  HPV16 | 4715 [1358 to 16368] | 10962 [3489 to 34438] | 7607 [1379 to 41972]
  HPV18 | 1418 [450 to 4473] | 3694 [1522 to 8964] | 946 [296 to 3026]

7. Secondary Outcome: Serum Antibody Response (Total IgG) - Geometric Mean Titer
Description: as for outcome 6
Time Frame: At Day 30 post challenge dose of Human Papillomavirus 9-Valent vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 6 | 6
antibody titer
  HPV6 | 4579 [1930 to 10865] | 7308 [4781 to 11172] | 7371 [3757 to 14460]
  HPV11 | 3234 [1016 to 10297] | 6637 [3810 to 11559] | 6271 [3309 to 11884]
  HPV16 | 25808 [10472 to 63603] | 32051 [18808 to 54618] | 12364 [2957 to 51689]
  HPV18 | 6363 [2371 to 17082] | 4985 [1737 to 14304] | 1813 [805 to 4082]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at Day 7 (+/-1) and Day 30 (+/-3) following booster dose.
Description: Provincially reportable and serious adverse events only were collected.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02968420/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02968420/SAP_001.pdf